CLINICAL TRIAL: NCT05507333
Title: An Open Labelled Study to Evaluate Clinical Performance of the Gedea Pessary in Adult Women With Vulvovaginal Candidiasis
Brief Title: Clinical Performance of the Gedea Pessary in Adult Women With Vulvovaginal Candidiasis
Acronym: EpHect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gedea Biotech AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL4
Record Dates: First submitted 2022-05-24; First posted 2022-08-18 (Actual); Results first posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Vulvovaginal Candidiasis
Keywords: Vaginal Yeast Infection; Candidiasis, vulvovaginal; Genital diseases, female; Vaginitis; Vulvovaginitis; Vaginal diseases
MeSH Terms: conditions — Candidiasis, Vulvovaginal; Genital Diseases, Female; Vaginitis; Vulvovaginitis; Vaginal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gedea pessary (Other): Gedea pessary administration
  Interventions: Device: pHyph generation II

INTERVENTIONS:
Device: pHyph generation II — Daily administration of the Gedea pessary during 6 days
  Other Names: Gedea pessary

SUMMARY:
This is a multi-centre, multi-national study to evaluate the clinical performance and safety of treatment with Gedea Pessary in adult women with confirmed vulvovaginal candidiasis (VVC).

The study population will consist of post-menarchal, pre-menopausal females, 18 years or older, seeking care for VVC symptoms. A total of 26 patients are planned to be included in the study. On Day 0 (Screening, Visit 1), eligible patients will undergo a gynaecological examination, including collection of composite vulvovaginal signs-and-symptoms (CVVS) score data, and vaginal samples. Patients will be provided with 6 doses of Gedea Pessary that will be self-administered as a daily treatment (Days 0 to 5).

Patients will visit the clinic on Day 7 (+2 days, Visit 2) for gynaecological examinations, including collection of CVVS data for the assessment of clinical cure and reporting of AEs and concomitant medications. On Day 14 (±2 days, Visit 3), patients that did not have a clinical and mycological cure Day 7 will re-visit the clinic for additional gynaecological examinations, including collection of CVVS data for the assessment of clinical cure. Rescue treatment will be offered during visits 2 and 3, if necessary. Patients will have a final telephone follow-up on Day 25 (±3 days, Visit 4), for for reporting of AEs, concomitant medications and potential menstruation onset. Vaginal sampling for culture and sequencing, as well as vaginal pH measurements will be performed at the clinic on Day 0, Day 7, and Day 14. On Day 25, patients will self-perform vaginal swabs at home for sequencing and vaginal culture. Patient questionnaires for assessing VVC symptoms, will be used during the treatment period (Days 0 to 5), 1 day after the treatment (Day 6) and on Days 11 and 25. Usability will be assessed on Day 7, also via the patient questionnaire. The patient questionnaire will be based on an electronic patient reported outcomes (ePRO) system, i.e. a mobile application (ViedocMe™).

ELIGIBILITY:
Inclusion Criteria:

1. Having decisional capacity and providing written informed consent.
2. Adult, post-menarchal, pre-menopausal women, aged 18 years or older
3. Diagnosis of VVC, defined as:

   * Having a white or creamy vaginal discharge
   * At least 2 of the following signs and symptoms of VVC that are characterised as at least moderate: itching, burning, irritation, oedema, erythema, or excoriation.
   * KOH or saline preparation from the inflamed vaginal mucosa or secretions revealing yeast forms (hyphae or pseudohyphae) or budding yeasts.
4. Negative urine pregnancy test at Screening.
5. Refrain from using any intravaginal products (i.e. contraceptive creams, gels, foams, sponges, lubricants, or tampons, etc.) until Day 14.
6. Refrain from sexual intercourse or use a condom until Day 7.
7. Signed informed consent and willing and able to comply with all study requirements.

Exclusion Criteria:

1. Patients with known or apparent signs of other infectious causes of vaginal infection (BV, Trichomonas vaginalis, Neisseria gonorrhoeae, Chlamydia trachomatis, Herpes simplex, or human papillomavirus) at Screening.
2. Patients who are pregnant or breastfeeding.
3. Patients who were treated for VVC within 14 days prior to Screening.
4. Patients who are currently receiving anti-fungal therapy unrelated to VVC or has taken anti-fungal therapy within 14 days prior to Screening.
5. Patients who have received an investigational drug in a clinical investigation within 30 days prior to Screening.
6. Known/previous allergy or hypersensitivity to any product constituent or fluconazole.
7. Any medical condition that in the Investigator's judgements would make the patient unsuitable for inclusion.
8. More than 3 previous VVC infections during the last 12 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-03-16 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helena Kopp-Kallner, MD PhD, Principal Investigator — Obstetrics & Gynecology, Danderyd Hospital
Locations (4):
- Sweden (4):
  - Carlanderska, Gothenburg
  - KS Huddinge, Stockholm
  - Danderyds sjukhus, Stockholm
  - CTC MTC, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor webpage — http://gedeabiotech.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Gedea Pessary: Gedea pessary administration
  Gedea pessary: Daily administration of the Gedea pessary for 6 consecutive days
Period: Overall Study
Arm/Group | Gedea Pessary
Started | 26 (Received study treatment)
Completed | 25
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Gedea Pessary
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.1 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African descent | 0
  Asian or Pacific Islander | 3
  Caucasian | 22
  Mixed/Multi-racial | 0
  Other, Central American | 1
Region of Enrollment [Number; unit: participants]
  Sweden | 26
Childbearing potential [Count of Participants; unit: Participants]
  No | 0
  Yes | 26
Number of vulvovaginal candidiasis infections during the last 12 months [Number; unit: participants]
  0 | 1
  1 | 12
  2 | 7
  3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Clinical Cure Rate at Day 7-14
Description: Clinical cure was defined as the absence of signs and symptoms of vulvovaginal candidiasis (VVC) in terms of having a composite vulvovaginal signs-and-symptoms (CVVS) score equal to or below 3, with no intercurrent events (concomitant anti-fungal therapy or other treatments related to VVC due to lack of clinical performance prior to CVVS evaluation for the primary endpoint definition, treatment discontinuation due to lack of clinical performance, or rescue medication prior to CVVS evaluation for the primary endpoint definition).
  Each of the following vulvovaginal signs and symptoms was individually scored using the scoring scale below. The CVVS score is the sum of the 6 individual scores.
  * Vulvovaginal signs: erythema, edema, or excoriation
  * Vulvovaginal symptoms: itching, burning, or irritation
  Scoring scale: each score was objectively defined as: 0 = none (absent), 1 = mild (slight), 2 = moderate (definitely present), 3= severe (marked, intense)
Time Frame: Day 7-14
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Gedea Pessary
Number analyzed (Participants) | 26
Participants
  Clinical cure - No | 10
  Clinical cure - Yes | 16
Statistical Analysis 1: Comparison: Gedea Pessary; It was assumed that the true clinical cure rate was 54% in the treatment group, therefore a sample size of 24 patients was needed to obtain 80% power to show that the one-sided 95% CI for the clinical cure rate was above 30%. A sample size of 26 was used to account for patients with missing data. Hypotheses for the primary endpoint: Null hypothesis: Clinical cure rate is less than or equal to 30%. Alternative hypothesis (one-sided): Clinical cure rate is above 30%; Test type: Other; Proportion of clinically cured patients = 0.62, 95% CI 2-sided [0.4073 to 0.7909] — The proportion of clinically cured patients at Day 7-14 was calculated and presented together with a two-sided 95% CI based on the Wilson score for the proportion of "Yes" with continuity correction

2. Secondary Outcome: Continued Clinical Response to Treatment at Day 25
Description: Defined as the proportion of patients clinically cured on Day 7-14 and thereafter responding "no" to the yes/no question, "Have the symptoms recurred?" via telephone on Day 25.
Time Frame: Day 25
Population: Day 25 Per Protocol Analysis Set - the subset of patients in the Full Analysis Set for whom no protocol deviation judged to impact the Day 25 analyses was reported or identified.
Measure: Count of Participants; unit: Participants
Arm/Group | Gedea Pessary
Number analyzed (Participants) | 13
Participants
  Continued clinical response to treatment at Day 25 - Yes | 11
  Continued clinical response to treatment at Day 25 - No | 2
Statistical Analysis 1: Comparison: Gedea Pessary; Test type: Other; Proportion with cont. clinical response = 0.85, 95% CI 2-sided [0.5366 to 0.9729] — The proportion of participants with continued clinical response at Day 25 ("Yes") was calculated and presented together with a two-sided 95% CI. The CI was based on the Wilson score for the proportion of "Yes" with a continuity correction

3. Secondary Outcome: Combined Clinical and Mycological Cure at Day 7-14
Description: The proportion of patients reporting clinical cure Day 7-14 according to the primary endpoint and mycological cure (culture negative for growth of Candida species).
Time Frame: Day 7-14
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Gedea Pessary
Number analyzed (Participants) | 26
Participants
  Clinical cure and mycological cure - No | 16
  Clinical cure and mycological cure - Yes | 10
Statistical Analysis 1: Comparison: Gedea Pessary; Test type: Other; Proportion with clin and mycol. cure = 0.38, 95% CI 2-sided [0.2091 to 0.5927] — The proportion of participants with clinical and mycological cure at Day 7-14 ("Yes") was calculated and presented with a 95% CI. The CI was based on the Wilson score for the proportion of participants with "Yes" with a continuity correction

4. Secondary Outcome: Mycological Cure at Day 7-14
Description: Defined as the proportion of patients having a mycological cure as assessed by vaginal culture at Day 7-14.
Time Frame: Day 7-14
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Gedea Pessary
Number analyzed (Participants) | 26
Participants
  Mycological cure - No | 12
  Mycological cure - Yes | 14
Statistical Analysis 1: Comparison: Gedea Pessary; Test type: Other; Proportion with mycological cure = 0.54, 95% CI 2-sided [0.3375 to 0.7286] — The proportion of participants with mycological cure at Day 7-14 ("Yes") was calculated and presented with a 95% CI. The CI was based on the Wilson score for the proportion of participants with "Yes" with a continuity correction

5. Secondary Outcome: Mycological Cure at Day 25
Description: Defined as the proportion of patients achieving mycological cure as assessed by vaginal culture at Day 25.
Time Frame: Day 25
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Gedea Pessary
Number analyzed (Participants) | 13
Participants
  Mycological cure - No | 3
  Mycological cure - Yes | 10
Statistical Analysis 1: Comparison: Gedea Pessary; Test type: Other; Proportion with mycological cure = 0.77, 95% CI 2-sided [0.4598 to 0.9384] — The proportion of participants with mycological cure at Day 25 ("Yes") was calculated and presented with a 95% CI. The CI was based on the Wilson score for the proportion of participants recorded as "Yes" with a continuity correction

6. Secondary Outcome: Absence of Candida Hyphae in the Wet Smear
Description: Proportion of patients having an absence of Candida hyphae in the wet smear at Day 7-14.
Time Frame: Day 7-14
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Gedea Pessary
Number analyzed (Participants) | 26
Participants
  "Absence of Candida hyphae in the wet smear" - No | 11
  "Absence of Candida hyphae in the wet smear" - Yes | 15
Statistical Analysis 1: Comparison: Gedea Pessary; Test type: Other; Proportion with absence of Candida = 0.58, 95% CI 2-sided [0.3719 to 0.7603] — The proportion of participants that did not show Candida hyphae in the wet smear (absence of/"Yes") at Day 7-14 was calculated and presented together with a 95% CI based on the Wilson score for the proportion of "Yes" with a continuity correction

7. Secondary Outcome: Change in the Composite Vulvovaginal Signs and Symptoms (CVVS) Score From Screening to Day 7-14
Description: Each of the following vulvovaginal signs and symptoms was individually scored using the scoring scale below. The CVVS score is the sum of the 6 individual scores. A lower CVVS score means fewer vulvovaginal signs and symptoms. Change from the score at screening to the score at Day 7-14 is presented.
  * Vulvovaginal signs: erythema, edema, or excoriation (Investigator-assessed)
  * Vulvovaginal symptoms: itching, burning, or irritation (Patient-assessed)
  Scoring scale: each score was objectively defined as: 0 = none (absent), 1 = mild (slight), 2 = moderate (definitely present), 3= severe (marked, intense)
Time Frame: From Screening to Day 7-14
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale (Total range 0-18)
Arm/Group | Gedea Pessary
Number analyzed (Participants) | 26
score on a scale (Total range 0-18)
  CVVS score - Screening | 7.46 (2.02)
  CVVS score - Day 7-14 | 2.96 (2.54)
Statistical Analysis 1: Comparison: Gedea Pessary; Test type: Other; Mean Difference (Net) = -4.5, 95% CI 2-sided [-5.77 to -3.23], Standard Deviation 3.15 — The mean change in the score for composite vulvovaginal signs and symptoms from Screening to Day 7-14 was calculated and presented together with a 95% CI

8. Secondary Outcome: Change in the Composite Vulvovaginal Signs and Symptoms (CVVS) Score From Screening to Day 7-14 - Proportions
Description: Proportion of patients having a reduction in composite vulvovaginal signs and symptoms (CVVS) score on Day 7-14 compared to screening. NB. If the patient used rescue medication between Day 7 and Day 14, Day 7 data was used.
  Each of the following vulvovaginal signs and symptoms was individually scored using the scoring scale below. The CVVS score is the sum of the 6 individual scores.
  * Vulvovaginal signs: erythema, edema, or excoriation
  * Vulvovaginal symptoms: itching, burning, or irritation
  Scoring scale: each score was objectively defined as: 0 = none (absent), 1 = mild (slight), 2 = moderate (definitely present), 3= severe (marked, intense)
Time Frame: From Screening to Day 7-14
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Gedea Pessary
Number analyzed (Participants) | 26
Participants
  Reduction in signs/symptoms -No | 3
  Reduction in signs/symptoms -Yes | 23
Statistical Analysis 1: Comparison: Gedea Pessary; Test type: Other; Proportion with reduction CVVS score = 0.88, 95% CI 2-sided [0.6872 to 0.9697] — The proportion of participants having a reduction in signs and symptoms (CVVS scores) on Day 7-14 vs. Screening was calculated and presented with a 95% CI based on the Wilson score for the prop. with "Yes" with a continuity correction

9. Secondary Outcome: Proportion of Patients Having a Reduction in the Sum of the 3 Vulvovaginal Symptoms Scores (Itching, Burning, and Irritation) Over Time Compared to Screening
Description: The number of participants reported as "Yes" for having a reduction in CVVS score compared to screening is presented.
  Each of the following vulvovaginal signs and symptoms was individually scored using the scoring scale below. A lower CVVS score means fewer vulvovaginal symptoms.
  • Vulvovaginal symptoms: itching, burning, or irritation
  Scoring scale: each score was objectively defined as: 0 = none (absent), 1 = mild (slight), 2 = moderate (definitely present), 3= severe (marked, intense).
  Please note that assessments at Day 0 refer to the evening assessment post-treatment.
Time Frame: Day 1-7, Day 11, Day 14, Day 25
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Gedea Pessary
Number analyzed (Participants) | 26
Participants
  Day 0 (post-treatment): number analyzed (Participants) | 20
  Day 0 (post-treatment) | 6
  Day 1: number analyzed (Participants) | 25
  Day 1 | 14
  Day 2: number analyzed (Participants) | 25
  Day 2 | 15
  Day 3: number analyzed (Participants) | 25
  Day 3 | 17
  Day 4: number analyzed (Participants) | 24
  Day 4 | 16
  Day 5: number analyzed (Participants) | 25
  Day 5 | 21
  Day 6: number analyzed (Participants) | 24
  Day 6 | 22
  Day 7: number analyzed (Participants) | 24
  Day 7 | 22
  Day 11: number analyzed (Participants) | 19
  Day 11 | 16
  Day 14: number analyzed (Participants) | 10
  Day 14 | 9
  Day 25: number analyzed (Participants) | 22
  Day 25 | 20

10. Secondary Outcome: Change in the Sum of the 3 Vulvovaginal Symptoms Scores (Itching, Burning, and Irritation) Over Time Compared to Screening
Description: Change in the sum of the 3 vulvovaginal symptoms scores (itching, burning, and irritation) on Days 1-7, Day 11, Day 14 and Day 25, compared to screening.
  Vulvovaginal symptoms were individually scored using the scoring scale below.
  • Vulvovaginal symptoms: itching, burning, or irritation
  Scoring scale: each score was objectively defined as 0 = none (absent), 1 = mild (slight), 2 = moderate (definitely present), 3= severe (marked, intense).
  Please note that assessments at Day 0 refer to the evening assessment post-treatment.
Time Frame: Day 1-7, Day 11, Day 14, Day 25
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gedea Pessary
Number analyzed (Participants) | 26
units on a scale
  Day 0 (post-treatment): number analyzed (Participants) | 20
  Day 0 (post-treatment) | -0.200 (1.28)
  Day 1: number analyzed (Participants) | 25
  Day 1 | -0.560 (1.92)
  Day 2: number analyzed (Participants) | 25
  Day 2 | -1.24 (1.94)
  Day 3: number analyzed (Participants) | 25
  Day 3 | -1.40 (2.31)
  Day 4: number analyzed (Participants) | 24
  Day 4 | -1.50 (2.45)
  Day 5: number analyzed (Participants) | 25
  Day 5 | -2.48 (1.90)
  Day 6: number analyzed (Participants) | 24
  Day 6 | -2.75 (1.96)
  Day 7: number analyzed (Participants) | 24
  Day 7 | -3.00 (2.19)
  Day 11: number analyzed (Participants) | 19
  Day 11 | -2.63 (2.36)
  Day 14: number analyzed (Participants) | 10
  Day 14 | -2.70 (2.16)
  Day 25: number analyzed (Participants) | 22
  Day 25 | -3.77 (2.54)

11. Secondary Outcome: Usability, Measured by Patient Questionnaire on Day 6.
Description: Response to the question "is the vaginal pessary easy to use?"
Time Frame: Day 6
Population: Full Analysis Set (26 patients, 25 patients responded to the question)
Measure: Count of Participants; unit: Participants
Arm/Group | Gedea Pessary
Number analyzed (Participants) | 25
Participants
  No | 3
  Yes | 22

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the first administration of the Gedea Pessary until the end-of-investigation visit (e.g., 25 days)
Arm/Group | Gedea Pessary
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 16/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gedea Pessary (N=26)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1)
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 2 (2)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 3 (3)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 3 (3)
Bacterial vaginosis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Anal pruritus (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Vulvovaginal pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-07-04): https://cdn.clinicaltrials.gov/large-docs/33/NCT05507333/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-25): https://cdn.clinicaltrials.gov/large-docs/33/NCT05507333/SAP_001.pdf